CLINICAL TRIAL: NCT02275494
Title: The Influence of Leg Length Discrepancy After Total Hip Arthroplasty on Function and Quality of Life
Acronym: BioHipLLD
Status: Completed | Type: Observational
Sponsor: Sundsvall Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Sarwar-2
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Osteoarthritis; Leg Length Difference; Hip Arthroplasty
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- shortening group: Shortening group where the operated leg was more than 5mm shorter compared with the contralateral side
  Interventions: Procedure: Total hip arthroplasty
- Restoration group: the restoration control group where the operated leg was within 5mm shortening and 9mm lengthening compared with the contralateral side
  Interventions: Procedure: Total hip arthroplasty
- Lengthening group: The lengthening group where the operated leg became more than 9mm longer compared with the contralateral side.
  Interventions: Procedure: Total hip arthroplasty

INTERVENTIONS:
Procedure: Total hip arthroplasty — Cemented or uncemented total hip arthroplasty. No other intervention than observing patients operated according to routine practise at an orthopaedic department.

SUMMARY:
Leg length discrepancy (LLD) is a complication of THA and may result in patient dissatisfaction, gait disorder, greater trochanter pain, low back pain. In the literature, LLD is reported to vary widely among studies e.g. 6 to 35 mm. However, the threshold at which a LLD is clinically important is still a matter of debate. The aim of this study was to determine the influence of non-corrected LLD after THA on patients' reported hip function and quality of life. This prospective cohort study was conducted at Sundsvall Teaching Hospital in Sweden after it was approved by the regional ethics committee at Umeå University (No. 07-052M and No. 12-287-32M). Between September 2010 and April 2013, all patients with unilateral primary osteoarthritis (OA) treated with THA were considered for inclusion. Informed consent was obtained from all patients. Patients with secondary OA, previous spinal, pelvic, or lower limb injuries or fractures were excluded.

The primary outcome measure was the Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index that measures functional outcome (ref). The secondary outcome measure was the EQ-5D and visual analogue scale (VAS) scale. Patients were assessed preoperatively and at follow-up at 1 year postoperatively. The posterolateral approach was used in all operations. LLD was measured on the postoperative x-rays. patients were divided into three groups: shortening group where the operated leg was more than 5mm shorter compared with the contralateral side, the restoration control group where the operated leg was within 5mm shortening and 9mm lengthening compared with the contralateral side, and the lengthening group where the operated leg became more than 9mm longer compared with the contralateral side.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral primary osteoarthritis (OA) treated with THA were considered for inclusion.

Exclusion Criteria:

* Secondary OA.
* Previous spinal, pelvic, or lower limb injuries or fractures.
* Bilateral coxarthrosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with unilateral primary osteoarthritis (OA) treated with THA at the orthopaedic department in Sundsvall, Sweden were considered for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2010-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
WOMAC | 12-15 months

SECONDARY OUTCOMES:
EQ-5D | 12-15 months
Visual analogue scale | 12-15 months

REFERENCES:
- [Background] Ogawa K, Kabata T, Maeda T, Kajino Y, Tsuchiya H. Accurate leg length measurement in total hip arthroplasty: a comparison of computer navigation and a simple manual measurement device. Clin Orthop Surg. 2014 Jun;6(2):153-8. doi: 10.4055/cios.2014.6.2.153. Epub 2014 May 16. PMID 24900895
- [Background] Whitehouse MR, Stefanovich-Lawbuary NS, Brunton LR, Blom AW. The impact of leg length discrepancy on patient satisfaction and functional outcome following total hip arthroplasty. J Arthroplasty. 2013 Sep;28(8):1408-14. doi: 10.1016/j.arth.2012.12.009. Epub 2013 Mar 16. PMID 23507069
- [Background] McWilliams AB, Grainger AJ, O'Connor PJ, Redmond AC, Stewart TD, Stone MH. A review of symptomatic leg length inequality following total hip arthroplasty. Hip Int. 2013 Jan-Feb;23(1):6-14. doi: 10.5301/HIP.2013.10631. PMID 23397200
- [Background] Bertz A, Indrekvam K, Ahmed M, Englund E, Sayed-Noor AS. Validity and reliability of preoperative templating in total hip arthroplasty using a digital templating system. Skeletal Radiol. 2012 Sep;41(10):1245-9. doi: 10.1007/s00256-012-1431-4. Epub 2012 May 16. PMID 22588597
- [Background] Plaass C, Clauss M, Ochsner PE, Ilchmann T. Influence of leg length discrepancy on clinical results after total hip arthroplasty--a prospective clinical trial. Hip Int. 2011 Jul-Aug;21(4):441-9. doi: 10.5301/HIP.2011.8575. PMID 21818744
- [Background] O'Brien S, Kernohan G, Fitzpatrick C, Hill J, Beverland D. Perception of imposed leg length inequality in normal subjects. Hip Int. 2010 Oct-Dec;20(4):505-11. doi: 10.1177/112070001002000414. PMID 21157756
- [Result] Mahmood SS, Mukka SS, Crnalic S, Sayed-Noor AS. The Influence of Leg Length Discrepancy after Total Hip Arthroplasty on Function and Quality of Life: A Prospective Cohort Study. J Arthroplasty. 2015 Sep;30(9):1638-42. doi: 10.1016/j.arth.2015.04.012. Epub 2015 Apr 11. PMID 25922312